CLINICAL TRIAL: NCT02685995
Title: Randomized Trial Comparing VectorFlow Tunneled Dialysis Catheter to Palindrome Tunneled Dialysis Catheter
Brief Title: VectorFlow Tunneled Dialysis Catheter (TDC) Versus Palindrome TDC
Acronym: TDC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Teleflex (Industry); Arrow International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 823055
Record Dates: First submitted 2016-01-15; First posted 2016-02-19 (Estimated); Results first posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-01

CONDITIONS: Renal Failure Chronic Requiring Hemodialysis; Chronic Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Palindrome TDC (Active Comparator): TDC insertion with Palindrome will be in accordance with its FDA-approved indication under moderate sedation or general anesthesia with local anesthesia using 1% lidocaine in per institutional protocol. Following TDC insertion, the catheter may be used immediately. The goal of HD is typically to achieve a target effective blood flow of 300mL/min within the first 3 hemodialysis sessions. The dialysis records from each of the first three HD sessions will be reviewed by the study coordinator for (A) Blood flow rate (QB), (B) Arterial and venous lumen pressures, (C) Kt/V, and (D) Urea reduction ratio (URR). Additionally, need and use of thrombolytic infusion (ie t-PA) (other than single dose injection) to restore or improve patency and/or need for catheter exchange.
  Interventions: Device: Palindrome TDC
- VectorFlow TDC (Active Comparator): TDC insertion with VectorFlow will be in accordance with its FDA-approved indication under moderate sedation or general anesthesia with local anesthesia using 1% lidocaine in per institutional protocol. Following TDC insertion, the catheter may be used immediately. The goal of HD is typically to achieve a target effective blood flow of 300mL/min within the first 3 hemodialysis sessions. The dialysis records from each of the first three HD sessions will be reviewed by the study coordinator for (A) Blood flow rate (QB), (B) Arterial and venous lumen pressures, (C) Kt/V, and (D) Urea reduction ratio (URR). Additionally, need and use of thrombolytic infusion (ie t-PA) (other than single dose injection) to restore or improve patency and/or need for catheter exchange.
  Interventions: Device: VectorFlow TDC

INTERVENTIONS:
Device: VectorFlow TDC — TDC insertion with VectorFlow will be in accordance with its FDA-approved indication under moderate sedation or general anesthesia with local anesthesia using 1% lidocaine in per institutional protocol. Following TDC insertion, the catheter may be used immediately. The goal of HD is typically to achieve a target effective blood flow of 300mL/min within the first 3 hemodialysis sessions. The dialysis records from each of the first three HD sessions will be reviewed by the study coordinator for (A) Blood flow rate (QB), (B) Arterial and venous lumen pressures, (C) Kt/V, and (D) Urea reduction ratio (URR). Additionally, need and use of thrombolytic infusion (ie t-PA) (other than single dose injection) to restore or improve patency and/or need for catheter exchange.
  Other Names: ARROW-Clark™ VectorFlow™ Hemodialysis Catheter
  Arms: VectorFlow TDC
Device: Palindrome TDC — TDC insertion with Palindrome will be in accordance with its FDA-approved indication under moderate sedation or general anesthesia with local anesthesia using 1% lidocaine in per institutional protocol. Following TDC insertion, the catheter may be used immediately. The goal of HD is typically to achieve a target effective blood flow of 300mL/min within the first 3 hemodialysis sessions. The dialysis records from each of the first three HD sessions will be reviewed by the study coordinator for (A) Blood flow rate (QB), (B) Arterial and venous lumen pressures, (C) Kt/V, and (D) Urea reduction ratio (URR). Additionally, need and use of thrombolytic infusion (ie t-PA) (other than single dose injection) to restore or improve patency and/or need for catheter exchange.
  Other Names: Palindrome™ Dialysis Catheter
  Arms: Palindrome TDC

SUMMARY:
Randomized two-arm study examining 90 day primary patency of two FDA-approved tunneled dialysis catheters.

DETAILED DESCRIPTION:
The VectorFlow tunneled dialysis catheter is a novel symmetrical tip design tunneled dialysis catheter which in pre-clinical testing and retrospective review has improved flow and patency compared to other dialysis catheter designs. This study will compare 90 day patency rates of newly inserted VF catheters to the Palindrome catheter both of which are FDA approved devices and will inserted as standard of care. The Palindrome catheter has been selected as the comparison device because it is also a symmetrical tip catheter design and prior studies by the manufacturer of this device suggests it has a lower occlusion rate and better flow compared to other catheter designs.

ELIGIBILITY:
Inclusion Criteria:

* End stage renal disease or acute renal failure requiring hemodialysis through a tunneled dialysis catheter
* Age >18, Age <80
* Capable of giving informed consent

Exclusion Criteria:

* Coagulopathy defined as international normalized ration (INR) >2 which cannot be corrected with fresh frozen plasma
* Platelet count <50,000/microliter, which cannot be corrected with platelet transfusion
* Active skin infections at site of TDC insertion
* Presence of bacteremia or infected AVG/AVF within 7 days prior to enrollment
* Neutropenia defined as absolute neutrophil count less then 1,700/microliter
* Known central venous stenosis
* Occlusion of bilateral external and internal jugular veins or bilateral brachiocephalic veins or stenosis of the superior vena cava
* Functioning surgical HD access (ie AVG/AVF) or AVG/AVF which is expected to be functional within 90 days of enrollment
* Inability to provide informed consent
* Pregnant or nursing women
* In the event a physician does not feel that either catheter would be appropriate for a subject, the subject will not be eligible to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Nadolski, MD, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Hospital of the Unviersity of Pennsylvania, Philadelphia, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Vectorlow Dialysis Catheter Product Information — http://www.teleflex.com/en/usa/productAreas/interventionalAccess/productGroups/chronic-hemodialysis/products/vector/

RESULTS

PARTICIPANT FLOW:
Groups:
- Palindrome TDC: TDC insertion with Palindrome will be in accordance with its FDA-approved indication under moderate sedation or general anesthesia with local anesthesia using 1% lidocaine in per institutional protocol.
- VectorFlow TDC: TDC insertion with VectorFlow will be in accordance with its FDA-approved indication under moderate sedation or general anesthesia with local anesthesia using 1% lidocaine in per institutional protocol.
Period: Overall Study
Arm/Group | Palindrome TDC | VectorFlow TDC
Started | 50 | 50
Completed | 49 | 49
Not Completed | 1 | 1
Not completed — Insertion of immediately puncturable graft. | 1 | 1

BASELINE CHARACTERISTICS:
Population: ESRD patients receiving tunneled dialysis catheters
Groups:
- Total: Total of all reporting groups
Arm/Group | Palindrome TDC | VectorFlow TDC | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57 [49 to 67] | 59 [46 to 69] | 58 [46 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 26 | 46
  Male | 30 | 24 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 50 | 50 | 100
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Primary Patency - Intervention-free Interval (Measured in Weeks)
Description: The primary study endpoint will be primary patency at 90 days following catheter insertion. Primary patency is defined as an HD catheter which provides adequate hemodialysis (flow >300mL/min) without need for additional interventions (ie TPA infusions or catheter exchange) to maintain flow or correct device failure.
Time Frame: 30, 60 and 90 days
Measure: Median (Standard Error); unit: percentage of primary patency
Arm/Group | Palindrome TDC | VectorFlow TDC
Number analyzed (Participants) | 49 | 49
percentage of primary patency
  30 Days | 89.1 (6.2) | 95.5 (3.3)
  60 Days | 79.4 (10.0) | 87.2 (7.3)
  90 days | 71.5 (12.6) | 80.6 (9.8)

ADVERSE EVENTS:
Time Frame: 90 days from enrollment
Description: No adverse events occurred in this study
Arm/Group | Palindrome TDC | VectorFlow TDC
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-08-10): https://cdn.clinicaltrials.gov/large-docs/95/NCT02685995/Prot_SAP_ICF_000.pdf